CLINICAL TRIAL: NCT03799926
Title: ZG-801 Phase II Trial - Exploratory Study of Efficacy and Safety on Patients With Hyperkalemia, and Long Term Safety Study -
Brief Title: Exploratory Study of ZG-801 for the Treatment of Hyperkalemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZG-801-01
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — patiromer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Stratum 1: 8.4 g patiromer (Experimental): Non-dialysis subjects with serum potassium 5.1 to < 6.0 mEq/L range at baseline
  Interventions: Drug: patiromer
- Stratum 1: 16.8 g patiromer (Experimental): Non-dialysis subjects with serum potassium 5.1 to < 6.0 mEq/L range at baseline
  Interventions: Drug: patiromer
- Stratum 1: placebo of 8.4 g patiromer (Experimental): Non-dialysis subjects with serum potassium 5.1 to < 6.0 mEq/L range at baseline
  Interventions: Drug: placebo
- Stratum 1: placebo of 16.8 g patiromer (Experimental): Non-dialysis subjects with serum potassium 5.1 to < 6.0 mEq/L range at baseline
  Interventions: Drug: placebo
- Stratum 2: 8.4 g patiromer (Experimental): Non-dialysis subjects with serum potassium 6.0 to < 6.5 mEq/L range at baseline
  Interventions: Drug: patiromer
- Stratum 2: 16.8 g patiromer (Experimental): Non-dialysis subjects with serum potassium 6.0 to < 6.5 mEq/L range at baseline
  Interventions: Drug: patiromer
- Stratum 3: 8.4 g patiromer (Experimental): Dialysis subjects with serum potassium 5.5 to < 6.5 mEq/L range at baseline
  Interventions: Drug: patiromer
- Stratum 3: 16.8 g patiromer (Experimental): Dialysis subjects with serum potassium 5.5 to < 6.5 mEq/L range at baseline
  Interventions: Drug: patiromer

INTERVENTIONS:
Drug: patiromer — Patiromer starting dose: 1 packet/day, orally, once daily. The dose of patiromer could be titrated based on subject's serum potassium response (stratum 1)
  Arms: Stratum 1: 8.4 g patiromer
Drug: patiromer — Patiromer starting dose: 2 packets/day, orally, once daily. The dose of patiromer could be titrated based on subject's serum potassium response (stratum 1)
  Arms: Stratum 1: 16.8 g patiromer
Drug: placebo — Placebo starting dose: 1 packet/day, orally, once daily. The dose of patiromer could be titrated based on subject's serum potassium response (stratum 1)
  Arms: Stratum 1: placebo of 8.4 g patiromer
Drug: placebo — Placebo starting dose: 2 packets/day, orally, once daily. The dose of patiromer could be titrated based on subject's serum potassium response (stratum 1)
  Arms: Stratum 1: placebo of 16.8 g patiromer
Drug: patiromer — Patiromer starting dose: 1 packet/day, orally, once daily. The dose of patiromer could be titrated based on subject's serum potassium response (stratum 2)
  Arms: Stratum 2: 8.4 g patiromer
Drug: patiromer — Patiromer starting dose: 2 packets/day, orally, once daily. The dose of patiromer could be titrated based on subject's serum potassium response (stratum 2)
  Arms: Stratum 2: 16.8 g patiromer
Drug: patiromer — Patiromer starting dose: 1 packet/day, orally, once daily. The dose of patiromer could be titrated based on subject's serum potassium response (stratum 3)
  Arms: Stratum 3: 8.4 g patiromer
Drug: patiromer — Patiromer starting dose: 2 packets/day, orally, once daily. The dose of patiromer could be titrated based on subject's serum potassium response (stratum 3)
  Arms: Stratum 3: 16.8 g patiromer

SUMMARY:
To investigate the efficacy of each ZG-801 starting dose and the titration algorithm of ZG-801 for the treatment of hyperkalemia in Japanese patients.

To evaluate the safety of ZG-801 for the chronic use (total over 52 weeks). In addition, to confirm the safety after the discontinuation of ZG-801 treatment on 1 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18 - 80
* Informed consent given
* Serum Potassium measurement at baseline is 5.1 to < 6.5 mEq/L (Non-dialysis patients or 5.5 to < 6.5 mEq/L (Dialysis patients)

Exclusion Criteria:

* Subjects with hospitalization for hyper- or hypoglycemia with Type 2 diabetes or for acute exacerbations of heart failure within the previous 3 months
* Subjects with severe heart failure, defined as NYHA (New York Heart Association) class IV
* Subjects with uncorrected hemodynamically significant primary vascular disease or uncontrolled or hemodynamically unstable arrhythmia
* Subjects with coronary artery bypass graft, percutaneous intervention, or major surgery including thoracic and cardiac, within the previous 3 months or anticipated need during study participation
* Subjects with heart, liver (only Dialysis patients), or kidney transplant recipient, or anticipated need for transplant during the study period
* Subjects with any of the significant cardiovascular or cerebrovascular events within the previous 2 months
* Subjects with a history of or current diagnosis of a severe swallowing disorder, moderate to severe gastroparesis, or history of bariatric surgery, bowel obstruction or severe gastrointestinal disorders or major gastrointestinal surgery
* Subjects who cannot use the oral concomitant medication to be separate 3 hours from ZG-801 medication
* Subjects suspected of transient high potassium levels, such as those caused only by dietary effects

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Change in serum potassium from baseline to 1 week after the start of administration in each group of starting dose | Baseline to week 1

SECONDARY OUTCOMES:
Change in serum potassium 4 weeks after the start of administration in each group of starting dose | Baseline to week 4
Proportion of subjects with a normalized serum potassium level at 4 weeks after the start of administration in each group of starting dose | Week 4
Incidence of adverse events | Over 52-week study period
Incidence of adverse drug reactions | Over 52-week study period

CONTACTS AND LOCATIONS:
Locations (1):
- Zeria Investigative Sites, Kanagawa, Japan